CLINICAL TRIAL: NCT03579576
Title: Demonstration Project on Assessment of Simplified Antiviral Treatment Strategy for Hepatitis C in Myanmar
Brief Title: Simplified Antiviral Treatment Strategy for Hepatitis C in Myanmar
Status: Completed | Type: Observational
Sponsor: Right to Care (Other)
Collaborators: Community Partners International (Other); Myanmar Liver Foundation (Other); Boston University (Other); University of California, Los Angeles (Other); Ministry of Health and Sports, Myanmar (Other Government)
Responsible Party: Sponsor
Other Study IDs: EQUIPHCV01-MY
Record Dates: First submitted 2018-06-24; First posted 2018-07-06 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C; Hepatitis B; HIV Infections
Keywords: PWID; MSM; HCV; HIV
MeSH Terms: conditions — Hepatitis C; Hepatitis B; HIV Infections | interventions — Sofosbuvir; velpatasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dry Blood spots ( DBS) will collected at baseline, 4, 8, 12 and 24 weeks for viral load and resistance testing will be determination where applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCV infected patients: All participants found HCV infected with or without HIV will be initiated treatment and followed up until 24 weeks ( 12 weeks after treatment)
  Interventions: Drug: sofosbuvir 400 mg/velpatasvir 100 mg (SOF/VEL) orally once daily for 12 weeks with or without weight-based ribavirin.

INTERVENTIONS:
Drug: sofosbuvir 400 mg/velpatasvir 100 mg (SOF/VEL) orally once daily for 12 weeks with or without weight-based ribavirin. — Direct Acting anti-HCV drugs given to all HCV infected participants at baseline.Those with Co-infections like HIV and or HBV will be given treatment as per national guidelines.

SUMMARY:
The project will evaluate cost and treatment outcomes of a simplified hepatitis C virus (HCV) testing, treatment and care model integrated with HIV testing and treatment among key affected populations including people who inject drugs (PWID) in Myanmar.

DETAILED DESCRIPTION:
Affected populations will be screened for HCV and HIV and treated with direct a fixed-dose combination of sofosbuvir 400 mg/velpatasvir 100 mg (SOF/VEL) orally once daily for 12 weeks with or without weight-based ribavirin. Before and after completion of the treatment course viral load assessments will be undertaken using low-cost laboratory monitoring for comparison to standard HCV viral load measurement. Up to 800 patients enrolled on treatment will be followed up at 4, 8, 12 and 24 weeks when Sustained Viral Load ( SVL) will be determined. Safety monitoring will be undertaken at applicable visits for those on Ribavirin and all adverse events will be reported based on Good Clinical Practice. In addition to assessing to assessing cost outcomes, the project will assess HCV treatment efficacy in terms of sustained virologic response at 12 weeks after end of HCV treatment (defined as undetected HCV RNA or less than lower limit of detection), compare the cost of low cost HCV viral assay platforms to standard of care, assess rates of ART initiation and virologic suppression of HIV-infected persons within the simplified HCV testing and treatment model and impact of HIV co-infection in participants on the HCV treatment outcome of sustained virologic response (SVR12). The project will be conducted 3 treatment sites in Yangon, Mandalay, and Kachin state in Myanmar.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness of participant to provide informed consent.
2. Men and women age 18 years.
3. Active HCV infection as defined by detectable serum or plasma HCV RNA at any time prior to study entry. Documentation may be obtained from medical records if available. NOTE: If no medical records on HCV infection are available, active HCV infection must be confirmed by a detectable HCV RNA PCR prior to project entry.
4. Allowed HCV treatment history:

   1. HCV treatment naïve defined as not having been previously treated for Hepatitis C infection with any medications approved for the treatment of HCV in any country.
   2. HCV treatment experienced with interferon with or without ribavirin only (no prior DAA treatment).
5. Chronic Hepatitis B status must be documented by hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), and hepatitis B core antibody (HBcAb) testing. Participants with positive HBsAg must be already on an active HBV regimen at study entry.
6. HIV-1 infection status must be documented as either absent or present, as defined below:

   1. Absence of HIV-1 infection, as documented by rapid HIV test or HIV-1 enzyme immunoassay (ELISA) test kit, within 60 days prior to entry.

      OR
   2. Presence of HIV-1 infection, documented by rapid HIV test or HIV-1 ELISA test kit at any time prior to entry.

      OR
   3. HIV-1 infection confirmed by medical documentation as participant is registered in care at AIDS Center and receiving or preparing to initiate ARV treatment.
7. HIV co-infected participants taking ART or planning to initiate ART, should be:

   1. Tolerating ART for at least 2 weeks without signs of needing to modify or discontinue the ART regimen before initiating HCV treatment.

      AND
   2. The ART regimen must be a regimen that can be co-administered with SOF/VEL.
8. Participants who are assigned to receive ribavirin as part of the treatment protocol must have hemoglobin ≥11.0 g/dL
9. For females of reproductive potential who will receive ribavirin, a negative urine pregnancy test (urine -HCG with a sensitivity of <25 mIU/mL) within 48 hours prior to project entry (HCV treatment initiation) must be documented.
10. Male and female participants who are able to impregnate or become pregnant (ie, of reproductive potential) and are participating in sexual activity that could lead to pregnancy must agree to practice contraception/birth control as indicated below or agree to not participate in a conception process while on treatment with ribavirin through at least 12 weeks post-treatment.
11. Life expectancy >12 months, in the opinion of the site investigator

Exclusion Criteria:

1. Child-Pugh Score corresponding to Class B or C (decompensated cirrhosis). This requires assessment for encephalopathy and ascites, as well as measurement of serum bilirubin, albumin, and international normalized ratio (prothrombin time).
2. Breastfeeding or pregnancy if patient will be receiving ribavirin.
3. Known allergy/sensitivity or any hypersensitivity to components of drug(s) or their formulation.
4. Acute tuberculosis (TB) infection. They will be followed and offered enrolment when they complete TB treatment.
5. Renal impairment defined as estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2 or end-stage renal disease receiving dialysis as treatment with SOF/VEL is contraindicated (https://www.mdcalc.com/mdrd-gfr-equation).
6. Unwilling to provide informed consent for participation in the project.
7. Prior treatment with any HCV Direct Acting Agents (DAA).
8. Unable or unwilling to adhere to the HCV treatment course and monitoring in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are key population including Female Sex Workers, Men who have sex with men and People Who Use InjecaAll HCV-infected men and women aged 18 years or older. The study population eligible for HCV treatment will be HCV treatment naïve or experienced (pegylated interferon [PegIFN] and ribavirin [RBV] only), HCV-infected men and women aged 18 years or older with HCV genotype 1, 2, 3, 4, 5 or 6, with or without HIV-1 co-infection. Participants with compensated cirrhosis (Child-Pugh Class A) and hepatitis B infection will be eligible for HCV treatment. Patients with decompensated liver cirrhosis (Child-Pugh Class B or C) or prior treatment with HCV DAAs will not be eligible for treatment.
Sampling Method: Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Estimated cost of HCV screening per patient screened and per case identified and the cost per successfully treated patient for HCV mono-infected and co-infected participants | Two years. This will be after data on Viral load response is complete.
  The average cost to the provider per patient achieving SVR12 will be estimated, as will the average cost per other outcomes achieved, such as per patient screened and per patient remaining in care by other specified endpoints, stratified by HIV status and by any other important patient or site characteristics that are identified as drivers of cost. The study will also estimate the average cost to "produce" a successful outcome (SVR12), which is the ratio of total costs for the intervention for the entire sample enrolled to the number of patients achieving the primary outcome. This latter estimate captures the costs incurred for patients who do not have successful outcomes and thus relates resource utilization to health outcomes.
Overall Sustained Viral load response (SVR12) across all groups of HCV genotype, fibrosis stage, HIV and HBV co-infection. | 24 weeks ( 12 weeks post treatment)
  This will be the main treatment outcome of all patients initiated on treatment. Baseline viral load is done at entry with treatment initiated for those positive and eligible. Patients initiated on treatment will be assessed for viral load response at 24 weeks ( 12 weeks post treatment). This will also help in development of Care cascade for HCV testing, treatment and SVR12 in key populations co-infected with HIV/HCV, HIV/HCV/HBV, HBV/HCV and HCV mono-infected.

SECONDARY OUTCOMES:
HCV genotype and subtype | At baseline
  HCV Genotype and subtypes will be determined at entry for all patients. Frequency of resistance associated substitutions (RAS) among participants registered for the project will also be determined.
Validity and reliability of Cepheid GeneXpert in monitoring SVR12 | Testing done at baseline and 24 weeks
  150 patients will be evaluated for HCV viral load at entry and exit ( SVR12) comparing cepheid Gene Xpert and Roche real time PCR ( Standard method)
HIV Viral load among HCV/HIV co-infected patients | HIV Viral load at 24 weeks ( 12 weeks post HCV treatment)
  HCV/HIV co-infected patients will either be on treatment at the time of HCV treatment initiation but those not on ART will be initiated and will assess rates of ART initiation and virologic suppression of HIV-infected persons within the simplified HCV testing and treatment model.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Sanne, MBBCH,FRCP, Study Chair — Right to Care; Khin Pyone Khi, MBBS,FRCP,PhD, Principal Investigator — Myanmar Liver Foundation; Charles Chasela, PhD, Study Director — Right to Care
Locations (3):
- Burma (3):
  - Waimaw, Kāchen, Kachin State
  - Myanmar Liver Foundation Clinic, Mandalay
  - Myanmar Liver Foundation Charity Clinic, Yangon